CLINICAL TRIAL: NCT01996293
Title: Pharmacokinetics of Lamotrigine in Pregnant and Postpartum Women With Bipolar Disorder
Brief Title: Pregnant Women Taking Lamictal for Bipolar Disorder
Acronym: PK-LAPB
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Crystal Clark, Associate Professor, Northwestern University
Other Study IDs: 00079810
Record Dates: First submitted 2013-11-15; First posted 2013-11-27 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Bipolar Disorder
Keywords: pregnant; bipolar; lamotrigine; lamictal; women; female
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine; Triazines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum specimen will be obtained to measure lamotrigine and estradiol levels. Standard of care labs will be obtained on every participant that is eligible and signs informed consent. Participants will not have more than 50 ml of blood drawn every 8 weeks. Participants will also have the option to have blood drawn for DNA banking.
  Participants in the study that elect to receive analgesia for pain related to labor and have a spinal-epidural at Northwestern University will have CSF stored and banked for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lamotrigine for Bipolar: antepartum and peripartum women taking lamotrigine for Bipolar Disorder
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — Lamotrigine will be observed in women who have already under the guidance of a physician decide to continue lamotrigine for the treatment of Bipolar Disorder
  Other Names: Lamictal, Lamiktal, Labileno, Triazines

SUMMARY:
This study seeks to examine how the dose of lamotrigine (Lamictal) should be adjusted during pregnancy for women with Bipolar Disorder. The investigators predict that the concentration of Lamictal in women's blood will decrease during pregnancy, and increase after postpartum. Because the concentration of the medication is likely to decrease during pregnancy, it is important for doctors to know how much they should increase a patient's dose in order to prevent worsening of Bipolar symptoms. In this study, the investigators will ask that participants complete up to five overnight visits to our clinical research unit where their blood will be drawn every couple of hours, through an IV catheter, to measure how the concentration of lamotrigine (Lamictal) changes over time. Participants will be compensated for their time.

DETAILED DESCRIPTION:
There is an increased risk of recurrence of Bipolar Disorder (BD) episodes or worsening symptoms in pregnancy after the discontinuation of mood stabilizers. Similarly, changes in medication concentration due to the physiological changes in pregnancy may effectively reduce the medication dose and thus its efficacy in pregnancy. Therapeutic dose monitoring has proven to have great utility in preventing seizure recurrence in women with epilepsy (WWE), specifically, dose monitoring of lamotrigine (LTG). Similar guidelines to that of women with epilepsy would benefit pregnant women with BD who are taking lamotrigine (LTG) in pregnancy. However, the pharmacokinetics as well as the utility of therapeutic dose monitoring of LTG in pregnant patients with Bipolar Disorder has not been well studied.

This study is an observational protocol to explore the longitudinal pharmacokinetics (PK) of LTG during pregnancy and postpartum in 10 women with Bipolar Disorder. The correlation between changes in bioavailability and level-to-dose (L/D) ratios and increases in symptoms of depression, mania and anxiety and recurrence of syndromal BD episodes that fulfill Diagnostic and Statistics Manual of Mental Disorders (IV) (DSM4) criteria will be investigated.

The primary aims of this study are 1.) To assess the impact of the dynamic physiology of pregnancy on the L/D ratio and bioavailability of LTG in women with BD. 2.) To evaluate the correlations between maternal and umbilical cord LTG serum levels. 3.) To explore the relationship between declining LTG L/D ratios during pregnancy, bioavailability and the increase in psychiatric symptoms and recurrence of syndromal BD. 4.) To explore the relationship between declining LTG L/D ratios during pregnancy, bioavailability and the recurrence of anxiety symptoms.

Additionally this study will evaluate correlations between estradiol levels and change in LTG L/D ratios during pregnancy. To optimize the research yield from this investigation, participants will have the option to allow banking of cerebrospinal (CSF) fluid and DNA for future analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* If Pregnant, equal to or less than 26 weeks
* English-speaking
* DSM-IV Bipolar Disorder, any subtype
* Able to provide informed consent
* Daily dosing of Lamictal

Exclusion Criteria:

* Active substance abuse within last 6 months and/or positive urine drug screen
* Active suicidality
* No obstetrical care
* Antiepileptic drugs that affect metabolism of LTG
* Medications in FDA categories F or X that are not antimanic drugs
* Liver or kidney disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited broadly from Northwestern clinical services including Internal Medicine, OB/GYN, Family Medicine, and Psychiatry, registries, and from the local Chicagoland community. Patients that sign consent, complete the evaluation and meet criteria for Bipolar Disorder, any subtype, will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Serum concentration/elimination | An average of every 10 weeks; Hours 0, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 20, 24, or 0, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 13.5, 14.5, and 16
  For patients on 1x day dosing, serum levels will be obtained beginning at time 0 and at hours, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 20, 24 and L/D ratio will be determined at each time point. This series of serum levels will be completed an average of every 10 weeks across pregnancy, and postpartum. For patients on 2x dosing, serum levels will be obtained at hours 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 13.5, 14.5, and 16 hours.

SECONDARY OUTCOMES:
Infant (umbilical cord)/Maternal ratio of LTG | 30 min
  Ratio of umbilical cord (infant) LTG serum level to maternal LTG serum level will be determined at delivery.
Scores on depression assessment, Inventory of Depression Symptomatology- Self Report (IDS-SR) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  To determine if there is a pattern of increasing scores on self-report depression assessment (IDS-SR) and declining L/D ratios. Increasing scores indicate worsening symptoms or depression episode recurrence.
Scores on mania assessment, Young Mania Reporting Scale (YMRS) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  To determine if there is a pattern of increasing scores on clinician administered mania assessment (YMRS) and declining L/D ratios.
Scores on anxiety scale, Generalized Anxiety Disorder (GAD-7) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.

OTHER OUTCOMES:
Percent increase in estradiol levels and their correlation to percent decrease in LTG L/D ratio | Estradiol levels will be examined an average of every 10 weeks from the time the participant enters the study, up to 12 weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal T Clark, MD, MSc, Principal Investigator — Associate Professor
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clark CT, Klein AM, Perel JM, Helsel J, Wisner KL. Lamotrigine dosing for pregnant patients with bipolar disorder. Am J Psychiatry. 2013 Nov;170(11):1240-7. doi: 10.1176/appi.ajp.2013.13010006. PMID 24185239